CLINICAL TRIAL: NCT04584710
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2a Study of RTB101 as COVID-19 Post-Exposure Prophylaxis in Adults Age ≥65 Years
Brief Title: A Phase 2 Study of RTB101 as COVID-19 Post-Exposure Prophylaxis in Older Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Restorbio Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RTB101-211; 3R01AG064802-02S1 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: Mechanistic Target of Rapamycin (mTOR); Virus
MeSH Terms: conditions — COVID-19; Hereditary Sensory and Autonomic Neuropathies; Virus Diseases | interventions — dactolisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg daily RTB101 (Experimental): RTB101
  TORC1 inhibitor
  Interventions: Drug: RTB101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTB101 — Oral RTB101 10 mg hard gelatin capsule once daily for 2 weeks
  Other Names: Dactolisib; BEZ235
  Arms: 10 mg daily RTB101
Drug: Placebo — Oral matching placebo once daily for 2 weeks
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
The proposed trial will obtain preliminary data on the feasibility of studying RTB101 as compared to placebo for COVID-19 post-exposure prophylaxis in adults age ≥ 65 years to inform the design of a subsequent pivotal trial.

DETAILED DESCRIPTION:
The RTB101-211 study is a Randomized, Double-Blind, Placebo-Controlled Phase 2a Study of RTB101 as COVID-19 Post-Exposure Prophylaxis in Asymptomatic Adults Age ≥65 Years who: have SARS-CoV-2 detected on a surveillance nasal or nasopharyngeal swab OR live in the same house or apartment as someone who has laboratory-confirmed symptomatic COVID-19. The study is designed to obtain study feasibility data for RTB101 in an unbiased fashion and will inform the design of a subsequent pivotal trial.

ELIGIBILITY:
1. Informed consent must be obtained from the subject before any assessment is performed.
2. Adults (male and female) aged 65 years and over who are asymptomatic but:

   1. have SARS-CoV-2 detected during surveillance nasal or nasopharyngeal swab testing OR
   2. live in the same house or apartment as someone who has laboratory-confirmed symptomatic COVID-19 .
3. Sexually active male subjects with a partner of child-bearing potential must be willing to wear a condom while on study drug and for 1 week after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men with a partner of child-bearing potential to prevent delivery of the drug via seminal fluid.
4. Subject must be able to understand and comply with the requirements of the study including having internet access and an email account, willingness to answer an eDiary questionnaire on a personal electronic device each night, and willingness to answer the telephone questionnaires twice weekly

Exclusion Criteria:

1. Any subject who self-reports:

   1. As a current smoker, or stopped smoking within the past 6 months.
   2. As a previous smoker with a ≥10 pack year smoking history.
   3. Has a household member who currently smokes in the house.
2. Subjects with a medical history of chronic obstructive pulmonary disease (COPD), emphysema or chronic bronchitis requiring active treatment with a prescription medication
3. The subject has already had symptoms consistent with COVID-19 at screening.
4. Subjects who require chronic supplemental oxygen therapy at screening.
5. Subjects with current evidence of an unstable medical disorder including an unstable respiratory disorder, gastrointestinal disorder (including Child-Pugh class B and C hepatic impairment), renal disorder or hematologic disorder (including active leukemia) for which they have had an exacerbation of symptoms within the past month, or are undergoing a change in treatment.
6. The following cardiac conditions:

   1. Unstable angina pectoris
   2. History of myocardial infarction (MI), coronary bypass surgery, or any percutaneous coronary intervention (PCI) within 6 months prior to Screening
   3. Congestive heart failure requiring active treatment with a prescription medication
   4. Unstable or life-threatening cardiac arrhythmia

   a. Chronic stable atrial fibrillation is allowed
7. Subjects with a history of systemic autoimmune diseases (e.g., lupus, inflammatory bowel disease, rheumatoid arthritis, etc.).

   a. Psoriasis confined to the skin and eczema are allowed
8. Subjects receiving immunosuppressive therapy including chronic use of supraphysiologic steroids such as prednisone >10 mg daily (however, inhaled corticosteroids and acute use of higher doses of prednisone to treat conditions such as exacerbation of asthma or other acute conditions are allowed).
9. Subjects with an immunodeficiency disease, including a history of a positive human immunodeficiency virus (HIV) test result.
10. Subjects with a history of gastric bypass surgery.
11. Subjects who require treatment with strong CYP3A4 or CYP1A2 inhibitors or inducers, or subjects who require treatment with digoxin.
12. Use of any other investigational medication or participation in any other investigational study within 5 half-lives of the investigational medication, or within 30 days, whichever is longer; or longer if required by local regulations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
To determine the length of time from date of receipt of a positive SARS-CoV2 test result to date of first dose of study drug in asymptomatic adults age ≥ 65 years | Beginning of randomization through Week 2
  The number of days from the date of receipt of a positive SARS-CoV-2 swab test result to the date of first dose of study drug in asymptomatic subjects who:
  * have SARS-CoV-2 detected on a surveillance nasal or nasopharyngeal swab OR
  * live in the same house or apartment as someone who has laboratory-confirmed symptomatic COVID-19

SECONDARY OUTCOMES:
To determine the feasibility of using an eDiary to assess study drug compliance in the study drug population | Beginning of randomization through Week 2
  Study drug compliance determined from the number of capsules of study drug taken by the subject based on data reported in an eDiary
To determine the feasibility of using an eDiary to assess study drug compliance in the study drug population | Beginning of randomization through Week 2
  Study drug compliance determined from the number of capsules of study drug taken by the subject based on data from twice weekly phone calls
To determine the feasibility of using an eDiary to assess study drug compliance in the study drug population | Beginning of randomization through Week 2
  Study drug compliance determined from the number of capsules of study drug taken by the subject based on a pill count done by phone when subjects complete study drug treatment
To determine the feasibility of using an eDiary to assess COVID-19 symptoms in the study population | From time of first dose through Week 3
  Incidence and severity of COVID-19 symptoms based on data reported in an eDiary
To determine the feasibility of using an eDiary to assess COVID-19 symptoms in the study population | From time of first dose through Week 3
  Incidence and severity of COVID-19 symptoms based on data from twice weekly phone calls
To assess the incidence of treatment-emergent of AEs and SAEs in subjects assigned to RTB101 as compared to placebo | From time of first dose through Week 3
  Safety and tolerability will be assessed by report of AE/SAEs from first dose of study drug through Week 3
To determine the percentage of subjects treated with RTB101 as compared to placebo who develop symptomatic laboratory-confirmed COVID-19 from first dose through Day 14 | From time of first dose through Week 2
  The percentage of subjects who have SARS-CoV-2 detected on nasal or nasopharyngeal swab and who develop 2 or more concurrent symptoms of COVID-19 from first dose of study drug through Day 14
To determine the percentage of subjects treated with RTB101 as compared to placebo who die from any cause from first dose of study drug through Day 14 and 21 | From time of first dose through Week 3
  The percentage of subjects who die from any cause from first dose of study drug through Day 14 and 21
To determine the percentage of subjects treated with RTB101 as compared to placebo who develop laboratory-confirmed COVID-19 from first dose through Day 14 and are subsequently hospitalized for any reason through Day 21 | From time of first dose through Week 3
  The percentage of subjects who develop laboratory-confirmed COVID-19 from first dose of study drug through Day 14 and are subsequently hospitalized for any reason through Day 21
To determine the percent of subjects treated with RTB101 or placebo who have laboratory-confirmed SARS-CoV-2 infection regardless of symptoms from first dose of study drug through Days 7, 14, 21. | From time of first dose through Week 3
  The percentage of subjects who have SARS-CoV-2 detected on nasal or nasopharyngeal swab regardless of symptoms from first dose of study drug through Day 7, 14, and 21 among subjects who are not SARS-CoV-2 positive at screening or baseline

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Restorbio Inc.
Locations (2):
- United States (2):
  - University of Connecticut, UConn Center on Aging, Farmington, Connecticut
  - Hebrew Senior Life, Marcus Institute for Aging Research, Roslindale, Massachusetts

IPD SHARING:
Plan to Share IPD: No